CLINICAL TRIAL: NCT01023282
Title: Randomised, Double-blind, Placebo-controlled Study Evaluating Safety and Tolerability of ACR325 in Parkinson's Disease Patients, With Evaluation of the Effect on Levodopa Induced Dyskinesias as a Secondary Measure
Brief Title: Safety and Tolerability Study Evaluating ACR325 in Parkinson's Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroSearch A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACR325C005
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-06

CONDITIONS: Parkinson's Disease; Tolerability
Keywords: Parkinson's disease; Levodopa; Dyskinesia; ACR325
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACR325 (Experimental)
  Interventions: Drug: ACR325
- Placebo (Placebo Comparator)
  Interventions: Drug: ACR325; Drug: Placebo

INTERVENTIONS:
Drug: ACR325 — Capsules, dose titration from 25 mg to 75 mg bid or matching placebo. Duration of dosing: 3 weeks
Drug: Placebo — Capsules, dose titration from 25 mg to 75 mg bid or matching placebo. Duration of dosing: 3 weeks
  Arms: Placebo

SUMMARY:
The study will evaluate the safety and tolerability of ACR325 in Parkinson disease patients and evaluate the effect on levodopa induced dyskinesias.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson"s disease according to the United Kingdom Parkinson's Disease Society brain bank diagnostic criteria
* Levodopa induced dyskinesia

Exclusion Criteria:

* Previous surgery for Parkinson's disease
* Any current or history of heart condition or increased pro-arrhythmic risk
* Severe or ongoing unstable medical condition

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Paracelsus-Elena-Klinik, Kassel, Hesse
  - Klinik für Neurologie, Philipps-Universität Marburg, Marburg, Hesse